CLINICAL TRIAL: NCT06631716
Title: Evaluation of the Effectiveness of Mechanically Assisted Sputum Excretion
Brief Title: To Assess the Effectiveness of Three Distinct Mechanical Assisted Sputum Evacuation Apparatuses in the Treatment of Patients With Mechanical Ventilation-induced Atelectasis
Acronym: EOTEOMASE
Status: Not yet recruiting | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2037-02
Record Dates: First submitted 2024-09-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Mechanical Ventilation; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CVT — During mechanical ventilation, patients with atelectasis confirmed by chest CT, chest X-ray or lung ultrasound should be treated with mechanical assisted sputum evacuation, and the mechanical assisted sputum evacuation equipment used is CVT.
Device: HFCWO — During mechanical ventilation, patients with atelectasis confirmed by chest CT, chest X-ray or lung ultrasound should be treated with mechanical assisted sputum evacuation, and the mechanical assisted sputum evacuation equipment used is HFCWO.
Device: MetaNeb — During mechanical ventilation, patients with atelectasis confirmed by chest CT, chest X-ray or lung ultrasound should be treated with mechanical assisted sputum evacuation, and the mechanical assisted sputum evacuation equipment used is MetaNeb.

SUMMARY:
Retention of airway secretions is a common clinical problem in patients with mechanical ventilation. Effective removal of airway secretions requires a balance between the production and removal of airway secretions through the mucociliary transport system. Effective removal of airway secretions is the basic measure to maintain airway patency and normal alveolar ventilation and oxygenation. At present, a variety of mechanical assisted expectoration devices have been used to remove airway secretions in critically ill patients, including The MetaNeb® System(MetaNeb), High Frequency Chest Wall Oscillation(HFCWO) and (Cycloid Vibration Therapy)CVT. However, there is still a lack of sufficient evidence to evaluate the clinical efficacy of these three different mechanical assisted expectoration devices in airway management of patients with mechanical ventilation. This study aims to observe the clinical efficacy of three different mechanical assisted sputum evacuation devices in airway management of patients with mechanical ventilation atelectasis, and to provide a basis for optimizing the airway management scheme of patients with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* patients who were diagnosed as obstructed airway secretion clearance and required mechanical sputum evacuation in Sir Run Run Shaw Hospital, Zhejiang University School of Medicine. Among them, patients using CVT were included in the CVT cohort, patients using Metaneb were included in the Metaneb cohort, and patients using high-frequency chest wall oscillation (HFCWO) were included in the high-frequency chest wall oscillation (HFCWO) cohort.
* voluntarily participated in this study and signed the informed consent. If the subjects were unable to read and sign the informed consent form due to incapacity or other reasons, their guardians were required to act for them during the informed consent process and sign the informed consent form. If the subjects were unable to read the informed consent form (e.g., illiterate subjects), witnesses were required to witness the informed consent process and sign the informed consent.
* Invasive mechanical ventilation ≥48 hours.
* Atelectasis was confirmed by chest CT, chest X-ray or lung ultrasound.

Exclusion Criteria:

* BMI≥40kg/m2.
* Severe spinal and thoracic deformity.
* Known or suspected diaphragmatic dysfunction such as phrenic nerve rupture, neuromuscular disease, etc.
* untreated tension pneumothorax.
* Active bleeding in the lung.
* Severe hemodynamic instability (increased dose of vasoactive drugs within 2 hours or MAP≤65mmHg).
* Severe other organ dysfunction was expected to result in short-term death (7 days) or palliative treatment.
* Other reasons considered by the medical team not suitable for treatment.
* Pregnancy status.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were more than 18 years old, with invasive mechanical ventilation for more than 48 hours and atelectasis confirmed by chest CT, chest X-ray or lung ultrasound in Sir Run Run Shaw Hospital, Zhejiang University School of Medicine were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
CT | From enrollment to the end of treatment at 5 days
  3D Slicer 5.0.3 software was used to import the chest CT data set, which consisted of 1.25mm thick continuous CT slices obtained by a multi-slice spiral CT scanner under a conventional dose protocol (120Kv,150mA, pitch 1.0), and then the ''Lung CT Segment'' extension program was used. The lung regions were segmented by manually marking 13 marker points. After marking, all the lung regions were visually displayed, and then the region range was manually corrected using the tools selected in the ''Segment editor''. The ''Lung CT Analyzer'' extension program was then used to quantify the lung zones of ''hyperventilation'', ''normal ventilation'', ''hypoventilation'', and ''no ventilation'', and the proportion of no ventilation areas was obtained by software analysis.

IPD SHARING:
Plan to Share IPD: No